CLINICAL TRIAL: NCT00656786
Title: A Phase 1, Multi-center, Randomized, Double-Blind, Placebo Controlled Study of the Safety, Tolerability, and Systemic Absorption of Menadione Topical Lotion as an Emergent and Pre-emergent Treatment for Epidermal-Growth-Factor-Receptor (EGFR) Inhibitor-Associated Rash
Brief Title: Safety, Tolerability and Systemic Absorption of Menadione Topical Lotion for Epidermal-Growth-Factor-Receptor (EGFR) Inhibitor-Associated Rash
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBS701
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: EGFR Inhibitor-associated Rash

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Subjects will be treated if, after starting treatment with an EGFRi, acute signs and symptoms of rash on the face/neck and/or upper chest emerge, that are suspected of being related to the EGFRi treatment.
  Interventions: Drug: Menadione Topical Lotion
- Group 2 (Experimental): Subjects will receive pre-emergent rash treatment starting 1 day prior to beginning EGFRi therapy
  Interventions: Drug: Menadione Topical Lotion

INTERVENTIONS:
Drug: Menadione Topical Lotion — Menadione Lotion will be applied topically twice a day; beginning when the rash appears during EGFRi therapy.
  Arms: Group 1
Drug: Menadione Topical Lotion — Menadione Lotion will be applied topically twice a day, starting 1 day before EGFRi therapy.
  Arms: Group 2

SUMMARY:
This is a clinical research study of an experimental new medication, Menadione Topical Lotion (MTL). The study lotion is experimental and has not been approved for public use. Hana Biosciences, Inc., the company that is developing MTL, is the sponsor of this study. EGFR inhibitors are used to treat non-small cell lung cancer (NSCLC), pancreatic cancer, colorectal cancer, breast cancer and head and neck cancer. One of the side effects of EFGR inhibitors is skin toxicities including an acneform skin rash.

This study is a Phase 1 study. The main purposes of this study are:

* Evaluate the safety and tolerability of Menadione Topical Lotion as an emergent and pre-emergent treatment for EGFR inhibitor-associated rash
* Evaluate the systemic absorption and bioavailability of Menadione Topical Lotion as an emergent and pre-emergent treatment for EGFR inhibitor-associated rash

It is planned that up to 24 patients undergoing EGFR inhibitor therapy will take part in this study at multiple clinical centers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years old;
2. Have been prescribed an approved EGFRI to treat cancer and expect to begin this treatment within 14 days (i.e., any EGFRI that is approved for the treatment of cancer at the time of subject enrollment);
3. For Group 1: Agree to return to clinic at Visit 3 or at first acute signs and symptoms of rash (papular and/or pustular eruptions and/or nodules) on the face/neck and/or upper chest that is suspected of being related to the EGFRI therapy within 21 days after starting EGFRI therapy;

   For Group 2: Expect to start EGFRI therapy one day after starting treatment with study lotion;
4. Have an Eastern Co-operative Oncology Group (ECOG) performance rating ≤ 2 (see Appendix 1);
5. Have a life expectancy of at least 4 months;
6. Males or non pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study. Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea, or at least 6 weeks following surgical menopause (bilateral oophorectomy);
7. Females of childbearing potential males with female sexual partners of childbearing potential must agree to use one of the following acceptable birth control methods:

   1. Surgically sterile (hysterectomy or bilateral oophorectomy);
   2. Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation). Documentation is required;
   3. Intrauterine device in place for at least 3 months;
   4. Double-barrier method (condom and diaphragm) with spermicide for at least 14 days prior to screening and through study completion;
   5. Stable hormonal contraceptive (oral, topical, vaginal or implanted//injected) for at least 3 months prior to study and through study completion;
   6. Abstinence;
   7. Single-barrier method for at least 14 days prior to screening and through study completion for vasectomized males or females with vasectomized partners;
8. Able to understand and provide signed informed consent;
9. Females of childbearing potential must have a negative serum β-human chorionic gonadotropin (hCG) pregnancy test at Visit 1 and negative urine β-hCG pregnancy test at Visit 3 (Group 1) or Visit 2 (Group 2).

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible for enrollment.

1. A skin examination reveals the presence of any active disease (e.g., eczema), tattoos or other problems, such as open lesions, that could make the application site unacceptable for study drug lotion application, located on the face/neck and/or upper chest that, in the Investigator's opinion, could confound the evaluation of the rash;
2. Any clinically significant safety laboratory or diagnostic results that, in the opinion of the Investigator, would place the subject at undue risk if the subject were to participate in the study;
3. Any clinically significant finding or concurrent clinical illness in the physical examination or medical history that, in the opinion of the Investigator, would place the subject at undue risk if the subject were to participate in the study;
4. Undergoing any current treatment for cancer other than the prescribed EGFRI that in the opinion of the Investigator, would place the subject at undue risk if the subject were to participate in the study;
5. Prior treatment with any other marketed or investigational EGFRI therapy within the 3 months prior to screening (Visit 1);
6. Treatment with topical antibiotics, topical steroids, and other topical treatments on the face/neck and upper chest within 14 days of first study lotion application;
7. Systemic use of steroids will be stopped at Visit 1 and not allowed during the course of the study;
8. Treatment with vitamin K supplements or multivitamins containing any form of vitamin K should be stopped at Visit 1;
9. Known hypersensitivity to menadione or similar compounds including any of the inactive ingredients;
10. Treatment with oral anticoagulant therapy (i.e., Warfarin);
11. Any subjects with prior history of bleeding and hematologic disorders;
12. Clinically significant abnormal laboratory values at screening, to include but not limited to the following hematologic, renal and liver function laboratory values:

    1. Hematologic function:

       * Hemoglobin < 9.0 gL/dL or < 10.0 g/dL for subjects receiving hematopoietic growth factors, such as darbopoeitin alfa or epoetin alfa
       * ANC < 1,500/mm3 (or < 1.5 ×109/L)
       * Platelet count < 100,000/mm3 (or < 100 ×109/L)
    2. Renal function:

       • Serum creatinine > 1.5 mg/dL or < 133 umol/L (SI units) or calculated estimated creatinine clearance < 60 ml/min/1.73 m2 based on Cockcroft and Gault formula
    3. Hepatic function:

       * Aspartate transaminase (AST) or alanine transaminase (ALT) > 3 × institutional upper limit of normal (ULN) or > 5 × institutional ULN if documented liver metastasis
       * Total bilirubin > 2 × institutional ULN or > 5 × institutional ULN if documented liver metastasis
13. Treatment with any cosmetic cream, make-up or products such as sun screen, oils, powders, perfumes, lotions, ointments, etc. to the anticipated study lotion application area within 3 days before treatment or during the treatment period;
14. Known or suspected pregnancy, lactation or planned pregnancy (females and males);
15. Clinically significant mental illness (to be determined by the Investigator);
16. Exposure to any investigational agent within 2 weeks or 3 half-lives prior to randomization (Visit 3, Day 1 for Group 1 or Visit 2, Day 1 for Group 2);
17. The subject will be disqualified if they have a rash for longer than 5 days at a grade of 3 or more prior to administration of first menadione dose (per CTCAE v3.0 terminology [see Appendix 2]);
18. Subject has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04-03 (Actual); Primary Completion 2009-12-30 (Actual); Study Completion 2009-12-30 (Actual)

PRIMARY OUTCOMES:
To evaluate safety, tolerability and systemic absorption of Menadione Topical Lotion as an emergent and pre-emergent treatment for EGFR inhibitor-associated rash | 6 weeks

SECONDARY OUTCOMES:
To evaluate skin rash status as an emergent and pre-emergent treatment for EGFR inhibitor-associated rash | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Colavincenzo, MD, Principal Investigator — Robert H. Lurie Cancer Center, Northwestern University; Vera Hirsh, MD, Principal Investigator — McGill University; Milan Anadkat, MD, Principal Investigator — Washington University School of Medicine; Serena Mraz, MD, Principal Investigator — Solano Clinical Research; Cliff Perlis, MD, Principal Investigator — Fox Chase Cancer Center, Rockledge, PA; Madeline Duvic, MD, Principal Investigator — MD Anderson Cancer Center, Houston, TX; Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (6):
  - Solano Clinical Research, Vallejo, California
  - Robert H. Lurie Cancer Center, Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Fox Chase Cancer Center, Rockledge, Pennsylvania
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- McGill University, Montreal, Quebec, Canada